CLINICAL TRIAL: NCT01358539
Title: Pain Education for Patients With Painful Bone Metastases Undergoing Palliative Radiotherapy: Reducing Pain by Increasing Patient's Knowledge and Self-management
Brief Title: Palliation: the Effect of Education on Pain
Acronym: PEEP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Kankerbestrijding (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ZonMW 11510007
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Bone Metastases
Keywords: palliation; pain education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pain education (Experimental): Patients receiving pain education
  Interventions: Behavioral: Pain education
- No Pain education (No Intervention): Control group, patients receiving no pain education

INTERVENTIONS:
Behavioral: Pain education — Patients receiving pain education
  Arms: Pain education

SUMMARY:
Rationale: Although radiotherapy is an effective palliative treatment for patients with painful bone metastases with over 70% responders, pain intensity is not always sufficiently controlled. Recent analyses from the randomized Dutch Bone Metastasis Study on 1157 patients show that during weekly follow up, 35% of the patients remain above a pain intensity level of 4 on a numeric rating scale (range 0-10) despite pain medication. According to the WHO criteria, a pain intensity of 5 or higher prompts treatment. As advised in the CBO guideline 'Pijn bij Kanker' educating patients can improve patient empowerment and thereby pain control. However, the effect of a nurse-led education of patients undergoing palliative radiotherapy for painful bone metastases has not been investigated yet.

Objective: This project investigates whether nurse-led pain education in addition to standard care results in better control of pain in patients referred for palliative radiotherapy.

Study design: A national multicenter phase 3 study (n=450).

Study population: Patients with painful bone metastases referred for short schedule radiotherapy.

Intervention: Patients will be randomized between standard care or standard care with the Pain Education Program, a nurse-led pain education. The pain Education Program will be provided on the same day the radiotherapeutic treatment will start. The nurse will first assess the knowledge of a patient based on a structured interview. Thereafter, lacunas will be taught using the 'Pijninstructie Programma' (Pain Education Program). In addition, nurses will telephone patients at regular intervals during follow-up to monitor their needs.

Main study parameters/endpoints: The primary outcome of this randomized multicenter study is a decrement of the number of patients whose worst pain intensity remains above 4 at any time during the 12 weeks of follow up with regard to the control group. The secondary outcome is improvement of quality of life.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: All patients will fill out the Brief Pain Inventory, the EORTC QLQ-C15-PAL and the EORTC QLQ-BM22 at baseline and, thereafter, weekly for 12 weeks after randomization.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* uncomplicated painful bone metastases
* primary malignancy is a solid tumour
* pain intensity on a numeric rating scale of 5 or higher
* indication for short-term radiotherapy
* able to fill out Dutch questionnaires
* able to follow instructions
* informed consent provided

Exclusion Criteria:

* Hematological malignancy
* Long-term schedule radiotherapy
* Life expectancy shorter than three months
* Karnofsky Performance Score of 40 or less

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2010-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
a decrement of the number of patients whose worst pain intensity remains above 4 | 12 weeks
  The primary outcome of this randomized multicenter study is a decrement of the number of patients whose worst pain intensity remains above 4 at any time during the 12 weeks of follow up with regard to the control group.

SECONDARY OUTCOMES:
improvement of quality of life | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: A KL Reyners, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands